CLINICAL TRIAL: NCT06649981
Title: Intestinal Microbiota Transplant as a Strategy to Enhance the Resilience Capacity of the Elderly Aiming to Retain Muscular, Cognitive, and Metabolic Functions in a Stressful Environment.
Brief Title: Aging Resilience Through Microbiota Optimization and Regulation
Acronym: ARMOR
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gonzalo Jorquera, PhD (Other)
Collaborators: Universidad de los Andes, Chile (Other)
Responsible Party: Sponsor-Investigator, Gonzalo Jorquera, PhD, Research director, University of Chile
Organization: University of Chile (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: WL-DR-GJ; Dynamic resilience programme (Other: Wellcome Leap)
Record Dates: First submitted 2024-10-14; First posted 2024-10-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Resilience; Cognitive Function and Well-Being; Muscle Function, Handgrip Strength Test; Insulin Sensitivity
Keywords: FMT; Resilience; gut microbiota; aging; cognition; muscle function; metabolic function
MeSH Terms: conditions — Insulin Resistance | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: Our research is structured as a randomized, placebo-controlled, double-blind clinical trial.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo group (Placebo Comparator): The first group receives a placebo (no FMT capsule)
  Interventions: Dietary Supplement: Placebo Capsule(s)
- FMT group (Experimental): The second group receives FMT from young-trained donors
  Interventions: Dietary Supplement: FMT capsule

INTERVENTIONS:
Dietary Supplement: FMT capsule — A lyophilized gut microbiota capsule derived from a rigorously screened, healthy, and physically active donor, free of gastrointestinal diseases, antibiotic use, and chronic conditions. The donor diverse microbiome is supported by a nutrient-rich diet and active lifestyle. The lyophilization process preserves microbial integrity, offering a high-potency dose aimed at restoring and optimizing the gut microbiome of older adults.
  This intervention is specifically designed for older adults to enhance resilience to stress, cognitive function, muscular strength, and metabolic health. It is part of a controlled clinical study with follow-up assessments at weeks 1, 4, 8, and 20 post-intervention. This targeted approach distinguishes it from other microbiome-based therapies by focusing on comprehensive health benefits for an aging population.
  Arms: FMT group
Dietary Supplement: Placebo Capsule(s) — A placebo capsule will be used in this study to serve as a control, allowing us to objectively assess the true effects of the lyophilized gut microbiota intervention. The use of a placebo is essential to eliminate bias and ensure that any observed outcomes can be confidently attributed to the actual intervention rather than to psychological or other non-specific effects.
  The placebo capsule will be identical in appearance, size, shape, and color to the interventional capsule to maintain blinding for both participants and researchers. This ensures that neither group knows which capsule is being administered, thereby preserving the study's integrity and validity by preventing any expectations or beliefs from influencing the results.
  Arms: Placebo group

SUMMARY:
Sarcopenia, characterized by the progressive loss of muscle mass and strength in older adults, is a key factor in health deterioration. It affects 15% of people between 65 and 80 years old and over 50% of those over 80, compromising autonomy and increasing the risk of diseases. Sarcopenia not only impacts muscle function but also bone health, mobility, and is associated with cardiometabolic diseases and cognitive decline.

It has been proposed that changes in the gut microbiota in aging individuals, known as gut dysbiosis, contribute to sarcopenia. Species diversity decreases, and bacterial representation is altered, which could impair muscle function through various pathways, such as mitochondrial dysfunction, chronic inflammation, and disruption of protein synthesis. Muscle function loss is strongly associated with cognitive and metabolic impairment in older adults.

Recently, it has been demonstrated that fecal microbiota transplantation (FMT) is an effective procedure for modulating gut microbiota and has proven highly effective in managing cases of Clostridium difficile-associated chronic diarrhea. The main objective of this project is to carry out FMT from young, physically active donors to a cohort of older adults to evaluate its effect on muscle, cognitive, and metabolic function.

Why donors who exercise? There is growing evidence that gut microbiota diversity is increased in young, physically active individuals. The FMT is planned to be administered through lyophilized microbiota capsules. By restoring microbial diversity, it is expected to improve the quality and function of skeletal muscles, leading to greater cognitive and metabolic resilience.

This project has great potential to develop an innovative approach for treating highly debilitating diseases that affect older adults, based on the lyophilization and encapsulation of gut microbiota from young, trained donors, which can be easily stored in a conventional freezer. Due to the high percentage of older adults worldwide and the high prevalence of sarcopenia within this age group, the aim of the project is to address a significant public health issue with a large target population eager for options to promote muscle health, functional autonomy, as well as cognitive and metabolic well-being.

DETAILED DESCRIPTION:
Skeletal muscle loss in old age is a critical point for the development of very serious health conditions affecting the quality of life of older adults, such as loss of autonomy, loss of healthy cognition, and the development of complex metabolic diseases. Additionally, intestinal microbiota can be modulated through fecal microbiota transplantation (FMT), and possibly this modulation could have direct effects that promote muscle health. Therefore, this project aims to investigate whether modifying the intestinal microbiota in older adults through FMT using young and trained donors can enhance skeletal muscle health and function, leading to greater resilience, reducing cognitive decline, and metabolic dysfunction associated with aging, especially in stressful contexts.

The donors would be young and trained individuals. Why trained donors? There is growing evidence that the composition of the intestinal microbiota is regulated by physical exercise. In animal studies, chronic exercise has been shown to increase the biodiversity of the intestinal microbiota and reduce systemic and intestinal inflammation. The bacterial profile associated with exercise is specific, for example, it does not correspond to that associated with a healthy diet, suggesting that physical activity allows for the development of a specific microbial profile in intestinal bacterial communities. Several studies have observed that changes in the intestinal microbiota associated with exercise are beneficial for promoting intestinal mucosal integrity and overall metabolic function in the individual.

In humans, intestinal bacterial biodiversity has been observed to be higher in athletes compared to sedentary subjects (normalized by body weight, age, and gender). In fact, there is evidence that a chronic exercise routine can restore the intestinal microbiota to a healthy profile in individuals with intestinal dysbiosis. In rats and mice, chronic exercise increases the biodiversity of Firmicutes, Bifidobacteria, and Actinobacteria and reduces the proportion of Bacteroides. Some data show how the presence of intestinal microbiota affects muscle performance, for example, it was found that germ-free mice had greater swimming endurance compared to germ-free mice, and when the latter were colonized with bacteria in the gut, the mice increased their physical endurance and swam for longer.

The main objective of this project is to carry out fecal microbiota transplants (FMT) from physically active young donors to a cohort of older individuals to evaluate their effect on muscle, cognitive, and metabolic function. FMT in older adults is planned to be performed by administering lyophilized microbiota capsules. By restoring microbial diversity, it is expected to improve the quality and function of skeletal muscles, leading to greater cognitive and metabolic resilience. It is important to mention that modifications of the intestinal microbiota have been associated with direct and specific effects on brain and metabolic functions, so the FMT from young and trained donors proposed in this project could have. This project has great potential to develop an innovative approach to treating highly debilitating diseases affecting older adults, based on the lyophilization and encapsulation of intestinal microbiota from young and trained donors, which can be easily preserved in a conventional freezer. This approach has been previously implemented for the treatment of C. difficile infection, with outstanding results. This idea will have a profound impact on the quality of life of adult and elderly patients, as it can be an alternative or complementary option to physical exercise therapy that older adults must undergo to prevent or treat sarcopenia, but often cannot be adequately achieved due to physical limitations associated with old age. Due to the high percentage of older adults worldwide and the high prevalence of sarcopenia among older adults, the researchers aim to address a significant public health issue with a large target population eager for options to promote muscle health, functional autonomy, as well as cognitive and metabolic well-being.

RESEARCH QUESTION. The hypothesis is as follows: Intestinal microbiota transplantation from young, trained donors promotes resilience through the enhancement of muscle function, thereby preserving cognitive and metabolic performance in older individuals exposed to stressful situations.

GENERAL AND SPECIFIC OBJECTIVES. General Objective To demonstrate that fecal microbiota transplantation from young and physically trained donors promotes muscle performance, preventing cognitive and metabolic decline in older individuals in a stressful context.

Specific Objectives To evaluate the effect of fecal microbiota transplantation (FMT) from trained young donors on the muscular health of aged individuals, correlating the results with the degree of stress exposure of the elderly recipients of FMT.

To assess the effect of fecal microbiota transplantation (FMT) from trained young donors on cognitive parameters of elderly recipients, correlating the results with individuals stress levels and modifications of muscle function after FMT.

To evaluate the effect of fecal microbiota transplantation (FMT) from trained young donors on metabolic parameters of elderly recipients, correlating the results with individiduals stress levels and modifications of muscle function after FMT.

In these objectives, researchers aim to investigate whether FMT from trained young donors can improve muscle function in older individuals, with beneficial consequences on cognitive and metabolic functions, correlating the results with the degree of stress exposure of the participants.

EXPERIMENTAL DESIGN. The research is structured as a randomized, placebo-controlled, double-blind clinical trial. Researchers will work with a group of 92 elderly individuals (aged 65-84 years, both women and men). All the characteristics mentioned in the experimental design, along with the fact that the researchers aim to evaluate the safety of the intervention and explore potential benefits of the treatment (FMT in this case) - such as muscular, cognitive, or metabolic improvements - in the context of a condition or disease (aging and a stressful environment), support the classification of this research as a Phase I clinical study. Participants will be recruited at Clínica Universidad de los Andes or the Institute of Nutrition and Food Technology (INTA) of the Universidad de Chile, after signing an informed consent document. FMT will be administered using capsules of lyophilized fecal microbiota manufactured at the Center for Biomedical Research and Innovation (CIIB) of the Universidad de los Andes.

Fecal Microbiota Donors. The donors will be young individuals (aged 20 to 35 years, 2 males and 2 females), physically active, who engage in at least 150 minutes of high-intensity aerobic physical activity per week, as this type of training improves the diversity and production of short-chain fatty acids (SCFAs) of the human intestinal microbiota. The Global Physical Activity Questionnaire (GPAQ) and actigraphs will be used to measure physical activity in donors 2 weeks before stool donation. For donor selection, individuals will be considered to have reached a metabolic equivalent (MET) of 600 minutes or more per week.

Donors will meet all criteria for donating fecal microbiota (criteria already established for FMT treatment in patients with CDAD.

During the initial stage of the selection process, the medical history and risk behavior of potential donors will be assessed using a specialized questionnaire. The questionnaire will be administered by a medical professional. Objective evaluation includes the consequences of a specific response for the selection process. The topics and elements to be addressed in this questionnaire are listed in Table 1.

TABLE 1. Elements to Evaluate During Donor Selection Prior to Approval for Fecal Microbiota Transplantation (FMT)

Infectious Diseases

* History of or exposure to infectious diseases with chronic activity: HIV, hepatitis B virus (HBV), hepatitis C virus (HCV), unsuccessfully eradicated Helicobacter pylori, syphilis, malaria, trypanosomiasis, tuberculosis, Chagas disease, strongyloidiasis.
* Any currently active or relevant infection within the last 6 months.
* Live attenuated virus vaccination within the last 8 weeks. Country of birth. Risk Behaviors
* Current or previous intravenous drug use.
* High-risk sexual behavior within the last 6 months.
* Travel to high-risk foreign countries within the last 6 months.
* Current occupation in an environment facilitating the acquisition of potential pathogens (e.g., veterinarian, animal caretaker, ranger, prison worker).
* Tattooing, piercing, or acupuncture within the last 6 months.
* Major surgery within the last 6 months.
* Contact with human blood (e.g., accident, needle stick injury) within the last 6 months.
* History of incarceration.
* Prior tissue/organ transplant.
* Blood product transfusion (e.g., packed red blood cells, plasma, platelets, immunoglobulins) within the last 6 months of medical history.

Medical History

* Chronic diseases.
* (Risk of) Creutzfeldt-Jakob disease.
* Allergies or atopy (e.g., food or drug allergies, asthma).
* Hospitalization within the last 4 months.
* Ongoing pregnancy.
* Antibiotic treatments, scheduled or received within the last 3 months.
* Regular medications or nutritional supplements.
* BMI (accepted if ≥20 and ≤25 kg/m2).
* Age (accepted if ≥18 and ≤30 years).

Intestinal Health

* Previous or scheduled gastrointestinal surgery, except for appendectomy.
* Gastrointestinal symptoms in the last 3 months (e.g., diarrhea, constipation, hematochezia, vomiting, abdominal pain), or adenomatous polyps or sessile serrated lesions (removed).
* Any other relevant clinical sign or symptom in the last 3 months (e.g., fever or rash).

In addition to all the infectious agents described in Table 2, SARS-CoV-2 will also be ruled out through RT-PCR in the stool. The presence of E. coli ST131 will be studied through classical culture and PCR typing, as well as the presence of antibiotic resistance genes. If positive results are obtained for these markers, the individual cannot be a donor. For each dose of FMT, a minimum of 150 grams of stool will be used, transported to the laboratory under the most anaerobic conditions possible (GutAlive system https://www.microviable.com/en/gutalive-2/) and in the shortest time possible from collection. Stool is a complex sample due to its variable water content, and the only way to standardize the dose is by the weight of the stool, as the amount of final powder can vary greatly. Therefore, the number of resulting capsules may vary widely. However, the microbial load will be equivalent as long as same logarithmic order is maintained. Stool will be lyophilized by mixing it with semi-skimmed lactose-free milk at a ratio of 1:2 as a cryoprotectant. The mixture will be homogenized in a Stomacher (230 rpm), solid residues will be removed by gentle centrifugation (500 rpm 5 min), and then all microorganisms will be collected by centrifugation (10,000 rpm 15 min). The supernatant will be removed, and the pellet will be frozen at -80°C for at least 1 hour, after which it will be lyophilized at -50°C for 18-20 hours. The obtained powder will be encapsulated in enteric-coated capsules in batches that will be stored in the absence of moisture at 4°C with a shelf life of 6 months. An aliquot of all processes will be stored at -80°C, and sample and donor traceability will be carried out with RedCap software.

Elderly Participants Number of participants: 92 Ethnicity : Chilean population. Chile has a population with homogeneous ethnicity, with indigenous (40%) and European (60%) ancestries.

Age: 65-84 years Biological sex: 46 males and 46 females

Study's recruitment, randomization, intervention, and follow-up process, organized in the following steps:

* Recruitment: Participants are recruited and undergo an eligibility evaluation. They are assessed to determine if they meet the inclusion criteria and do not meet the exclusion criteria.
* Informed Consent: Eligible participants who meet the study criteria provide their informed consent to participate.
* Pre-intervention Evaluations: Before the intervention, participants are assessed to classify them based on their levels of stress and anxiety.
* Randomization: A total of 92 participants are randomized into 2 groups:

Placebo group (n=46) IMT group (n=46)

Intervention: Participants in the four groups undergo the assigned intervention:

The first group receives a placebo capsule The second group receives IMT capsule (Intervention of Interest)

Follow-up: Follow-up evaluations are conducted at weeks 1, 4, 8, and 20 post-intervention for all groups to assess the outcomes of the interventions.

This research is structured as a randomized, placebo-controlled, double-blind clinical trial. This structure allows the study to compare the effects of the intervention (IMT) versus a placebo across different stress level classifications.

Pre-Intervention Assessments:

The 14-item Perceived Stress Scale (PSS-14) will be used to assess the level of stress in participants. Depressive symptoms will be evaluated using the 15-item Geriatric Depression Scale (GDS), which assesses mood disorder symptoms commonly associated with depression experienced in older adults (both documents attached). Anxiety symptoms will be measured using the Beck Anxiety Inventory (BAI), which is designed to obtain a measure of anxiety that is relatively independent of depression (attached). These instruments have high reliability and validity in community samples, which will allow us to classify our volunteers into low stress-anxiety and medium/high stress-anxiety groups. A post hoc analysis will be conducted to evaluate the effects of IMT on participants with low and medium/high stress levels.

To favor the establishment of the new ecosystem, the intestinal microbiota density of the participants will be reduced before the FMT with rifaximin (a suitable non-absorbable antibiotic for intestinal decontamination) for 3 days, 1,200 mg/day, administered in 2 daily doses. The antibiotic and its administration schedule will be provided to the participants.

The FMT will be conducted in the Clinical Trials Unit of the Universidad de los Andes Clinic by administering 4 capsules (containing a compact lyophilized preparation) prepared from approximately 150 grams of feces. Control subjects will receive placebo capsules with identical appearance to the capsules containing the intestinal microbiota lyophilized material. Free transportation will be provided to the participants between their homes and the Universidad de los Andes Clinic.

Researchers will conduct this study using only non-invasive tests and analyses. All proposed assessments to measure muscle, cognitive, and metabolic functions will be carried out before and after the FMT (from 1 to 20 weeks after the FMT). These assessments will be conducted at the Ambulatory Care Health Center of the National Institute of Agricultural Technology (CEDINTA). Free transportation will be provided to the participants between their homes and the CEDINTA. All participants will undergo medical history before and after the intervention to obtain information about overall health status, medication use, antibiotics, and dietary supplements, history of intestinal diseases, and any other intestinal disorder that may alter the intestinal microbiota.

Researchers will calculate the Frailty Index (FI) in participants from all groups before and after the FMT. The FI will be assessed using a combined method of clinical and laboratory parameters. Firstly, researchers will use a self-reported FI created with 30 variables to assess health status. Variables comprise different types of health problems, including diseases (n=9), symptoms (n=6), disabilities for living (n=6), psychological problems (n=2), Romberg test, physical performance, Geriatric Depression Scale (GDS) score, and Mini-Mental State Examination (MMSE) score. For binary variables, the presence of an impairment will be coded as "1"; and its absence as "0". For each three-level variable, 0.5 will be used to represent an intermediate response level. For the MMSE, it will be coded as 0 if >23, 0.5 if MMSE=15-23, and 1 if MMSE≤14, while GDS will be recoded as 0 if GDS<11) and 1 if GDS≥11. Secondly, a laboratory-based FI (FI-lab) will identify 15 parameters based on 9 laboratory tests, in addition to pulse, systolic and diastolic blood pressure, pulse pressure, BMI, and waist circumference. A normal reference range will be used to compare each parameter, where "0" indicates values within the normal range and "1" indicates values outside the reference range. Finally, researchers will combine the two FIs to construct a 45-item FI (FI-combined). Each FI-combined will be defined as the score of each parameter of an individual divided by the total number of parameters considered, with the FI ranging from a theoretical minimum of 0 (no impaired parameters present) to a maximum possible of 1.0 (all impaired parameters present).

For the assessment of muscle sarcopenia, researchers will measure lean and fat mass using dual-energy X-ray absorptiometry (DEXA) and creatinine excretion. A standard dynamometer will be used to measure isometric strength. Additionally, the Short Physical Performance Battery and the 6-minute walk test will be applied to estimate maximum oxygen consumption. Physical activity will be evaluated using an actigraph for 7 days. Researchers will measure the thickness of the rectus femoris muscle and the muscle pennation angle in the participants' thighs using ultrasound. As biomarkers for sarcopenia, creatine kinase (CK), skeletal muscle troponin T (sTnT), insulin-like growth factor-1 (IGF-1), C-reactive protein, vitamin D, TNF-α, IL-6, IL-1β will be measured in blood.

For cognitive performance, participants will be assessed on a set of higher cognitive abilities such as attention, executive functions, working memory, language, and processing speed, among others, before and after the FMT intervention. The Montreal Cognitive Assessment (MoCA), Trail Making Test A and B, Digit Span Forward and Backward, Frontal Assessment Battery (FAB), and Verbal Fluency (FAS) will be administered (attachments). Participants' quality of life will be assessed using the SF-36 questionnaire, one of the most commonly used and evaluated instruments for Health-Related Quality of Life (HRQoL).

For metabolic function, a comprehensive analysis of metabolic markers in blood such as insulin, glucose, total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, and transaminases (ALT, AST, gGT) will be performed in fasting conditions. Researchers will study the presence of non-alcoholic fatty liver disease (NAFLD) using ultrasound imaging. Additionally, concentrations of metalloproteinases-9 and IL-6 in serum will be measured by ELISA, as these markers have been proposed to be correlated with the severity of NAFLD in humans. Non-invasive scores of hepatic fibrosis will also be applied.

With the bacterial genomic DNA isolated from the fecal samples of the participants, researchers will study the microbiota profile using shotgun metagenomics or 16S gene sequencing. Samples will be collected from both young donors and older recipients before and after the FMT. Using bioinformatics tools, researchers will identify a bacterial signature in older adults who received FMT from trained young donors. Researchers will determine if this microbiome signature correlates with muscular, cognitive, and metabolic resilience, especially in the group experiencing higher stress. Researchers propose that key elements in this modified intestinal microbiota in older adults will serve as appropriate biomarkers for muscular, cognitive, and metabolic resilience in the context of aging.

SAFETY IMT performed by qualified personnel has not been associated with any serious adverse events, but mild or common adverse reactions may occur. Marcella et al. (2021) analyzed the presence of adverse reactions to IMT in a systematic review, evaluating 129 studies involving 4,241 patients. They found that the most common adverse effects were transient diarrhea (10%), transient abdominal cramps/discomfort (7%), nausea, and vomiting (<5%) within 24 hours post-IMT. Transient fever, abdominal distension, fatigue, and borborygmi have also been reported in less than 2% of cases. Constipation (2%) and excess flatulence (3%) were reported during follow-up.

Severe adverse reactions, such as bacteremia and death as a direct consequence of IMT, are extremely rare (incidence <0.1%) and occurred only in patients with diseases causing damage to the digestive mucosa. These diseases (inflammatory bowel disease, Crohn's disease, Clostridium difficile infection (CDI), and ulcerative colitis) are exclusion criteria for this study. Another study in 2022 evaluated the safety associated with the use of IMT in 5,344 patients affected by CDI. The researchers found that, overall, the safety profile was favorable in a medically complex patient population that usually has poor clinical outcomes. Among the cohort, 194 patients (3.6%) experienced one or more serious adverse reactions (SARs). SARs were more common among patients with severe or severe-complicated CDI (n = 94 [48.5%]). Among the SARs, six events (0.1%) were possibly related to IMT, all in patients who were severely immunocompromised. This included two patients with fever, as well as one with abdominal pain in a patient with severe-complicated CDI and breast cancer. Additionally, two patients developed systemic inflammatory response syndrome-one after a heart transplant and one after a kidney transplant. There was one reported case of an inflammatory bowel disease (IBD) flare-up in a patient with a history of ulcerative colitis not controlled with biological therapy and immunomodulators. None of the reported SARs were definitively related to IMT. Notably, no cases of sepsis or transmission of infectious diseases related to IMT, including infections with multi-drug-resistant organisms, were reported. This study will not include patients with CDI or those who are severely immunocompromised.

Finally, another systematic review and meta-analysis in 2022 searched for IMT studies in patients with CDI, using the rate of SARs related to IMT as the primary outcome. Secondary outcomes included SARs unrelated to IMT and minor adverse events associated with IMT. The combined analysis of 5,099 patients who received 5,551 IMTs showed that SARs related to IMT developed in less than 1% of patients. The combined rate of SARs unrelated to IMT was higher, reaching 2.9%. The combined rate of minor adverse events also showed infrequent self-limited gastrointestinal and systemic discomfort. This meta-analysis supports IMT as a safe option for treating recurrent CDI.

For IMT performed exclusively in the elderly population, a study of 31 patients with an average age of 77 years with CDI reported that 87% of patients resolved their infection, and the most common adverse event reported in 4 (13%) of 31 respondents was the subjective worsening of arthritis. Another study that performed IMT on 35 elderly patients (average age 77 years) with CDI reported no serious adverse effects.

In summary, the international experience using IMT reported in the literature shows the high safety of this procedure. However, the following risks should be considered: (1) Infection: Although IMT has been screened for pathogenic bacteria, viruses, fungi, and parasites, there is a risk of transmitting known and unknown infectious organisms contained in the donor's stool. There is also a theoretical risk of bacterial overgrowth in the small intestine. Rarely, bacteremia (e.g., E. coli, Klebsiella), sepsis, and fatal events can occur after IMT; (2) Exacerbation of inflammatory bowel disease (IBD) in individuals with underlying IBD; (3) Allergy/anaphylaxis to antigens present in the donor's stool; (4) Transmission of non-infectious diseases: There is a theoretical risk of developing diseases that may be related to the donor's gut microbiota. These include obesity, metabolic syndrome, cardiovascular diseases, autoimmune conditions, allergic/atopic disorders, neurological disorders, psychiatric conditions, and malignancies. This risk is very limited in the study, as individuals with these known conditions are excluded from stool donation according to the donor screening procedures explained in this protocol.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65-84 years
* Men and women
* Involuntary total body weight variation in the last 6 months < 10%
* Self-sufficiency (with a score >60 on the Barthel index)
* Fasting plasma glucose ≤ 7.2 mmol/l or glycosylated hemoglobin (HbA1c) ≤ 8% in the last 6 months.
* Must be able to swallow capsules

Exclusion Criteria:

* Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg at selection
* Allergy to rifaximin
* Acute infection or inflammatory condition in the last 4 weeks
* Use of antibiotics in the last 12 weeks
* Use of probiotics in the last 12 weeks
* Hospitalization in the last 12 weeks
* Current or within the last 6 months use of insulin
* Difficulty swallowing (dysphagia)
* Diagnosis of Inflammatory bowel disease
* Diagnosis of Crohn's disease
* Diagnosis of Ulcerative colitis
* Diagnosis of Clostridium difficile infection
* Diagnosis of Colon cancer
* Treatment with immunosuppressive therapy for organ transplant
* Diagnosis of leukemia
* Diagnosis of lymphoma
* Diagnosis of mesenchymal diseases except osteoarthritis
* Corticosteroid users
* Biological therapy users
* Individuals with a history of autoimmune or chronic inflammatory conditions (rheumatoid arthritis, chronic or active hepatitis B or C, human immunodeficiency virus, pancreatitis, or liver cirrhosis)
* Individuals with an active malignancy,
* Current drug or alcohol abuse (more than three drinks per day or more than seven drinks per week).
* Diagnosis of dementia (To assess the presence of this disease at the time of enrollment, the following questions will be asked:

Have you been diagnosed with dementia? ___Yes ___ No Do you take any of these medications?

* Donepezil ___Yes ___No
* Rivastigmine ___Yes ___No If the answer is positive to any of these questions, the patient will be excluded from the study. If there are doubts about the cognitive status of the potential participant by the recruiter, a Mini-Mental State Examination (MMSE) will be conducted, and the score must be ≥ 20)

Ages: 65 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Isometric strength | Before and after FMT (4-20 weeks follow-up)
  A standard dynamometer will be used to measure isometric strength.
Functional Autonomy: Global Index of the Latin American Group for Maturity (GDLAM) | Before and after FMT (4-20 weeks follow-up)
  The Global Index of the Latin American Group for Maturity (GDLAM) will be used to assess three aspects of mobility: balance, gait speed, and lower limb strength for standing up from a chair
Adverse effects after FMT registration | after FMT (4-20 weeks follow-up)
  Incidence of adverse effects after FMT will be recorded (serious and non-serious reactions) for safety and tolerability evaluation.

SECONDARY OUTCOMES:
Frailty index (FI) | Before and after FMT (4-20 weeks follow-up)
  Researchers will calculate the Frailty Index (FI) in participants before and after FMT, using clinical and laboratory data. A self-reported FI will be created with 30 variables, including diseases, symptoms, disabilities, psychological issues, and performance tests, while a lab-based FI will assess 15 parameters from 9 tests. The two FIs will be combined into a 45-item FI, with scores ranging from 0 (no impairments) to 1.0 (all parameters impaired), to evaluate participants' overall health status.
Lean and fat mass content | Before and after FMT (4-20 weeks follow-up)
  Researchers will measure lean and fat mass using dualenergy X-ray absorptiometry (DEXA).
Gut microbiota composition | Before and after FMT (4-20 weeks follow-up)
  With the bacterial genomic DNA isolated from the fecal samples of the participants, we will study the microbiota profile using shotgun metagenomics or 16S gene sequencing. Samples will be collected from both young donors and older recipients before and after the FMT. Using bioinformatics tools, we will identify a bacterial signature in older adults who received FMT from trained young donors. We will determine if this microbiome signature correlates with muscular, cognitive, and metabolic resilience, especially in the group experiencing higher stress. We propose that key elements in this modified intestinal microbiota in older adults will serve as appropriate biomarkers for muscular, cognitive, and metabolic resilience in the context of aging.
Metabolic function evaluation | Before and after FMT (4-20 weeks follow-up)
  For metabolic function, a comprehensive analysis of metabolic markers in blood such as insulin, glucose, total cholesterol, LDL-cholesterol, HDL-cholesterol, triglycerides, and transaminases (ALT, AST, gGT) will be performed in fasting conditions.
Working memory evaluation | Before and after FMT (4-20 weeks follow-up)
  The Digit Span Forward and Backward tests will be used to assess aspects of working memory, attention, and short-term memory. The Digit Span Forward and Backward tests are scored by the number of correctly recalled sequences. Higher scores indicate better working memory and attention.
Cognitive funcion evaluation | Before and after FMT (4-20 weeks follow-up)
  The Trail Making Test (TMT) consisting of two parts, A and B, will be used to assess cognitive function, particularly attention, processing speed, mental flexibility, and executive function. The Trail Making Test (TMT) has two parts: TMT-A and TMT-B, both measured in seconds to complete. Lower times indicate better performance. Longer times suggest cognitive impairment, particularly in processing speed (TMT-A) and mental flexibility/executive function (TMT-B).
Mild cognitive impairment detection | Before and after FMT (4-20 weeks follow-up)
  The Montreal Cognitive Assessment (MoCA) will be used to detect mild cognitive impairment and assess various cognitive domains, such as attention, concentration, executive functions, memory, language, visuospatial abilities, and orientation. The Montreal Cognitive Assessment (MoCA) is scored from 0 to 30, with higher scores indicating better cognitive function. A score of 26 or above is considered normal, while lower scores suggest increasing cognitive impairment.
Creatinine excretion | Before and after FMT (4-20 weeks follow-up)
  Creatinine levels in 24h urine will be evaluated
Physical activity | Before and after FMT (4-20 weeks follow-up)
  Physical activity will be evaluated using an actigraph for 7 days
Thickness of the rectus femoris muscle and the muscle pennation angle | Before and after FMT (4-20 weeks follow-up)
  Thickness of the rectus femoris muscle and the muscle pennation angle will be measured in the participants' thighs using ultrasound.
Evaluation of sarcopenia biomarkers in blood | Before and after FMT (4-20 weeks follow-up)
  As biomarkers for sarcopenia, creatine kinase (CK), skeletal muscle troponin T (sTnT), insulin-like growth factor-1 (IGF-1), C-reactive protein, vitamin D, TNF-α, IL-6, IL-1β will be measured in blood.
Frontal lobes of the brain function | Before and after FMT (4-20 weeks follow-up)
  The Frontal Assessment Battery (FAB) is a brief neuropsychological test designed to assess functions related to the frontal lobes of the brain and it will be used in the participants. The frontal lobes are involved in many higher cognitive functions, including executive function, decision-making, problem-solving, and control of behavior. The Frontal Assessment Battery (FAB) is scored from 0 to 18, with higher scores indicating better frontal lobe function. Lower scores suggest greater impairment in executive functions, such as abstract thinking, mental flexibility, and inhibitory control.
Phonemic fluency evaluation | Before and after FMT (4-20 weeks follow-up)
  The Verbal Fluency (FAS) test will be used to measure a person's ability to generate words under certain constraints, often used to evaluate executive function, language, and cognitive flexibility. The Verbal Fluency (FAS) test is scored based on the number of words generated within 60 seconds for each letter (F, A, S). Higher scores indicate better verbal retrieval and executive function, while lower scores suggest potential impairments in language or cognitive flexibility. There is no strict maximum score, but performance is compared to normative data based on age and education.
Quality of life evaluation | Before and after FMT (4-20 weeks follow-up)
  Participants' quality of life will be assessed using the SF-36 questionnaire. The SF-36 questionnaire assesses quality of life across 8 domains, each scored from 0 to 100, with higher scores indicating better health. It provides summary scores for physical and mental health.
NAFLD evaluation | Before and after FMT (4-20 weeks follow-up)
  The presence of non-alcoholic fatty liver disease (NAFLD) will be studied using ultrasound imaging.
NAFLD biomarkers in blood | Before and after FMT (4-20 weeks follow-up)
  Concentrations of metalloproteinases-9 and IL-6 in serum will be measured by ELISA, as these markers have been proposed to be correlated with the severity of NAFLD in humans.
Hepatic fibrosis evaluation | Before and after FMT (4-20 weeks follow-up)
  Non-invasive scores of hepatic fibrosis will also be applied. The FIB-4 index is a non-invasive score used to estimate liver fibrosis based on age, AST, ALT, and platelet count. It helps assess the degree of liver scarring, particularly in conditions like NAFLD. The FIB-4 score helps categorize the degree of liver fibrosis:
  Score < 1.45: Suggests minimal or no fibrosis (low risk). Score between 1.45 and 3.25: Suggests significant fibrosis (intermediate risk) Score > 3.25: Suggests advanced fibrosis or cirrhosis (high risk).

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Jorquera, PhD, Study Director — University of Chile; Ricardo Espinoza, MD, Principal Investigator — Universidad de Los Andes
Locations (2):
- Chile (2):
  - Clínica Universidad de los Andes, Santiago, Santiago Metropolitan
  - INTA - Universidad de Chile, Santiago, Santiago Metropolitan